CLINICAL TRIAL: NCT05115357
Title: Efficacy of Ultrasound-Guided Pecto-Intercostal Fascial Block Versus Transversus Thoracic Muscle Plane Block for Postoperative Analgesia in Cardiac Surgery
Brief Title: Pecto-Intercostal Fascial Block Versus Transversus Thoracic Muscle Plane Block in Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Abdullah Nabeih Abdullah Eloraby, Assistant lecturer of Anesthesiology and Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34494/2/21
Record Dates: First submitted 2021-11-03; First posted 2021-11-10 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Pecto-Intercostal Fascial Block; Transversus Thoracis Muscle Plane Block; Cardiac Surgery; Postoperative Analgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous analgesia group (No Intervention): Patients will receive systemic intravenous analgesia only.
- Pecto-Intercostal Fascial Block (PIFB) group (Experimental): Patients will receive PIFB on each side with an injection of 19 mL of 0.25% bupivacaine plus 1 ml of 4 mg dexamethasone.
  Interventions: Procedure: Pecto-Intercostal Fascial Block
- Transversus Thoracis Muscle Plane Block (TTP) group (Experimental): Patients will receive TTP on each side with an injection of 19 mL of 0.25% bupivacaine plus 1 ml of 4 mg dexamethasone.
  Interventions: Procedure: Transversus Thoracis Muscle Plane Block

INTERVENTIONS:
Procedure: Pecto-Intercostal Fascial Block — A high-frequency (7-12 Mhz) linear ultrasound transducer will be placed approximately 2 cm lateral to sternal edge in the 4th or 5th intercostal space. A 22-gauge, 50-mm needle will be inserted in-plane under ultrasound guidance. The needle will be advanced through the pectoralis major muscle, and the drug will be deposited in the pecto-intercostal fascial plane located between the pectoralis major muscle and the external intercostal muscles. The separation of the fascial plane and the spread of the drug could be observed on the ultrasound image .The procedure will be repeated on the other side of sternotomy to achieve bilateral blockade.
  Arms: Pecto-Intercostal Fascial Block (PIFB) group
Procedure: Transversus Thoracis Muscle Plane Block — The ultrasound probe will be placed in the longitudinal plane 1 cm lateral to the sterna border. the T4-T5 intercostal space will be identified under US. A parasternal sagittal view of the internal intercostal muscle and the transverses thoracis muscle between the 4th and 5th rib will be visualized above the pleura. A 22-gauge, 50-mm needle will be inserted inplane until the tip of the needle is located in the transversus thoracis muscle plane between the internal intercostal and transversus thoracis muscles . After excluding intravascular and intrapleural placement, local anesthetic will be administered in 5mL aliquots with intermittent aspiration.
  Arms: Transversus Thoracis Muscle Plane Block (TTP) group

SUMMARY:
The aim of this study is to compare the effect of Ultrasound-Guided Pecto-Intercostal Fascial Block versus Transversus Thoracis Muscle Plane Block on Postoperative Pain Analgesia in Cardiac Surgery

DETAILED DESCRIPTION:
Perioperative pain management is an essential component of the enhanced recovery pathway in patients undergoing cardiac surgery. The incidence of severe acute postoperative pain after median sternotomy is as high as 49%.

ELIGIBILITY:
Inclusion Criteria:

* 90 adult patients of both sexes aged (21-60) scheduled for cardio-pulmonary bypass cardiac surgery (valve replacement) with midline sternotomy

Exclusion Criteria:

* Patients' refusal.
* Cognitive impairment.
* History of drug abuse& chronic analgesic use
* History of allergy to local anesthetics.
* Emergency surgery
* Pre-existing major organ dysfunction including hepatic or renal failure, pulmonary insufficiency and left ventricular ejection fraction < 30%
* Known coagulopathy

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-12-24 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain score | 24 hours postoperative
  After extubation, patients will be evaluated for pain using numeric rating scale (NRS) score at 0,3,6,12,24 h for pain that ranged from (0 = no pain) to (10 = the worst imaginable pain). If score is ≥ 4, rescue analgesia will be given in the form of fentanyl in a dose of 0.5µg/kg by iv route.

SECONDARY OUTCOMES:
Total opioid consumption in first 24 hours after cardiac surgery | 24 hours Postoperative
  If the pain score is ≥ 4, rescue analgesia will be given in the form of fentanyl in a dose of 0.5µg/kg by iv route. The time to the first request for analgesia and the total fentanyl dose will be documented.
duration of mechanical ventilation | 24 hours Postoperative
  Duration of mechanical ventilation in intensive care unit.
Incidence of complications | 24 hours Postoperative
  Incidence of complications within 24hrs will be recorded as hematoma, pneumothorax and toxicity from local anathesitic.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The date will be available under a reasonable request of the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the end of the study